CLINICAL TRIAL: NCT01167595
Title: A Multicenter, Cluster Randomized Trial of Enhanced Protein-Energy Provision Via the Enteral Route Feeding Protocol in Critically Ill Patients: The PEP uP Protocol
Brief Title: Enhanced Protein-Energy Provision Via the Enteral Route in Critically Ill Patients
Acronym: PEPuP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinical Evaluation Research Unit at Kingston General Hospital (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Daren K. Heyland, Dr. Daren Heyland, Clinical Evaluation Research Unit at Kingston General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PEPuP cRCT
Record Dates: First submitted 2010-07-20; First posted 2010-07-22 (Estimated); Results first posted 2021-04-06 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Critically Ill
Keywords: Critically ill; Nutrition therapy; Enteral nutrition
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PEP uP Protocol (Experimental): PEP-uP protocol and treatment algorithm implemented for all patients in ICU.
  Interventions: Other: PEP uP Protocol
- Standard Feeding Protocol (No Intervention): Enteral feeds are guided by a standard feeding protocol specified by pre-printed ICU admission orders. The admitting physician has the option of initiating the enteral feeding protocol or keeping the patient nil per os (NPO).

INTERVENTIONS:
Other: PEP uP Protocol — Protocol documents (i.e. pre-printed order, algorithm for advancing feed, and algorithm for calculating rate of administering feed as per 24hour volume) and a slide presentation coupled with educational reminders (posters and bedside notices) and practice helps (tool to remind nurse to measure and report nutritional adequacy) will be made available to all nurses, in bedside manuals and/or on the local intranet.
  Arms: PEP uP Protocol

SUMMARY:
Critically ill patients are consistently underfed. Feeding protocols are standardized system tools used to guide nutrition practices, but to date have failed to improve delivery of nutrition. The PEP uP Protocol is a new enhanced feeding protocol. Twenty North American Intensive Care Units (ICUs) will assess baseline nutrition practices. Ten ICUs will be randomized to implement the PEP uP Protocol and educational intervention, and ten will be randomized to continue usual care. Nutrition practices will be reevaluated 6 months after baseline. The investigators hypothesize that the PEP uP Protocol will increase delivery of nutrition, and may ultimately lead to improved survival of critical illness.

DETAILED DESCRIPTION:
There is a well known and well described relationship between malnutrition, immune dysfunction, and infection. Critically ill patients are often hypermetabolic and can rapidly become nutritionally compromised. Repeated efforts over the past few years have not significantly improved the amount of calories delivered via the enteral route. Historically, feeding protocols have been used to guide the delivery of enteral nutrition (EN) but they frequently utilize conservative, reactionary approaches to optimizing nutrition.

We propose a new, innovative approach that protocolizes an aggressive set of strategies to providing EN and shifts the paradigm from reactionary to proactive followed by de-escalation if nutrition therapy is not needed. The key components of this new protocol are the following: 1) Starting feeds at the target rate based on increasing evidence that some patients tolerate starting nutrition at a higher rate of delivery and that slow start ups are not necessary. For patients who are hemodynamically stable, we propose to shift from an hourly rate target goal to a 24 hour volume goal and give nurses guidance on how to make up this volume if there was an interruption for non-gastrointestinal reasons. This 'volume-based' goal represents a significant shift in practice from traditional fixed hourly rate goals to a new protocol in which nurses can increase the hourly rate depending on how many hours they have left in the day to ensure that the patient receives the 24 hour volume within the day. 2) For patients who are deemed unsuitable for high volume intragastric feeds, we provide an option to initiate 'trophic feeds.' Trophic feeds represent an idea to provide a low volume of a concentrated feeding solution for 24 hours or longer, designed to maintain gastrointestinal structure and function rather than meet their protein and caloric goals. This option should reduce the numbers of patients ordered to be kept nil per os (NPO). Thus, PEP uP patients may gain some of the benefit of early EN. 3) To optimize tolerance in the early phase of critical illness, we propose to use a semi elemental feeding solution instead of a standard polymeric solution. There is some evidence that these semi elemental solutions are better assimilated than polymeric solutions in the critical care setting. These solutions can be changed to a more traditional polymeric solution once the patient is tolerating adequate amounts of nutrition. 4) Rather than wait for a protein debt to accumulate because of inadequate delivery of EN, protein supplements are prescribed at initiation of EN and can be discontinued if EN is well tolerated and they are receiving all their protein requirements through their standard EN. This strategy guarantees that the patient will most likely receive all their protein requirements in the early phase of their critical illness. 5) Rather than wait for a problem with gastrointestinal tolerance to develop, we propose to start motility agents at the same time EN is started with a re-evaluation in the days following to see if it is necessary. By preventing delayed gastric emptying, which frequently occurs in this patient population, we can improve nutritional adequacy. 6) Based on emerging evidence that a higher gastric residual volume (the volume of feeds remaining in the stomach when the bedside nurse aspirates the feeding tube) is safe and perhaps results in greater nutritional adequacy, we will include a higher gastric residual volume of 300ml in our protocol. It has been shown in one randomized trial that a feeding protocol that starts a motility agent empirically at the time of initiation of feeds and uses a higher threshold for a critical gastric residual volume (250 ml) improves nutritional adequacy.

Since the bedside nurses initiate and utilize feeding protocols to achieve target goals, we will couple this newer generational feeding protocol with a comprehensive nurse-directed nutritional educational intervention that will focus on its safe and effective implementation. This focus on nursing nutrition education represents a major shift away from traditional education which has focused on dietitians and physicians.

Our hypothesis is that this aggressive feeding protocol combined with a nurse-directed nutrition educational intervention will be safe, acceptable, and effectively increase protein and energy delivery to critically ill patients. We postulate that this increased provision of calories and protein may translate into improved clinical outcomes, particularly for the patients at the extremes of weight, but the current study is not powered to demonstrate such a difference.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adults (i.e. >18 years of age)
* Mechanically ventilated before or within the first 6 hours of admission to ICU

Exclusion Criteria:

* Nutrition (either EN or Parenteral Nutrition (PN)) started before admission to ICU
* Not intubated within 6 hours of admission to ICU
* Receiving non-invasive ventilation (i.e. mask ventilation) during the first 6 hours of ICU stay
* Moribund (as evidenced by death within 48 hours of admission to ICU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1059 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daren K Heyland, MD, Principal Investigator — Clinical Evaluation Research Unit
Locations (18):
- United States (9):
  - Phoenix Veterans Affairs Health Care System, Phoenix, Arizona
  - Medical Center of the Rockies, Loveland, Colorado
  - Washington Health Center, Washington D.C., District of Columbia
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - CoxHealth, Springfield, Missouri
  - Lakes Region General Hospital, Laconia, New Hampshire
  - Nassau University Medical Center, East Meadow, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - South Texas Veterans Health Care System Audie L. Murphy Division, San Antonio, Texas
- Canada (9):
  - Foothills Medical Centre, Calgary, Alberta
  - St Paul's Hospital, Vancouver, British Columbia
  - Rouge Valley Health System - Ajax and Pickering Site, Ajax, Ontario
  - William Osler Health Centre - Brampton Civic Campus, Brampton, Ontario
  - William Osler Health Centre - Etobicoke Campus, Etobicoke, Ontario
  - St Joseph's Healthcare, Hamilton, Ontario
  - The Credit Valley Hospital, Mississauga, Ontario
  - Rouge Valley Health System - Centenary Site, Scarborough Village, Ontario
  - Pasqua Hospital, Regina, Saskatchewan

REFERENCES:
- [Background] Heyland DK, Cahill NE, Dhaliwal R, Wang M, Day AG, Alenzi A, Aris F, Muscedere J, Drover JW, McClave SA. Enhanced protein-energy provision via the enteral route in critically ill patients: a single center feasibility trial of the PEP uP protocol. Crit Care. 2010;14(2):R78. doi: 10.1186/cc8991. Epub 2010 Apr 29. PMID 20429886
- [Result] Heyland DK, Dhaliwal R, Lemieux M, Wang M, Day AG. Implementing the PEP uP Protocol in Critical Care Units in Canada: Results of a Multicenter, Quality Improvement Study. JPEN J Parenter Enteral Nutr. 2015 Aug;39(6):698-706. doi: 10.1177/0148607114531787. Epub 2014 Apr 18. PMID 24748597
- See also: website — http://www.criticalcarenutrition.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted a cluster randomized trial of 18 ICUs in North America. Randomizing ICUs rather than individual patients was necessary to minimize the contamination of patients randomized to the usual care group who might have received care that was guided by the PEP uP protocol if it were operational in the same ICU at the same time
Units Other Than Participants: hospitals
Period: Overall Study
Arm/Group | PEP uP Protocol | Standard Feeding Protocol
Started | 522; 9 hospitals | 537; 9 hospitals
Completed | 522; 9 hospitals | 537; 9 hospitals
Not Completed | 0; 0 hospitals | 0; 0 hospitals

BASELINE CHARACTERISTICS:
Units Other Than Participants: ICUs
Groups:
- Total: Total of all reporting groups
Arm/Group | PEP uP Protocol | Standard Feeding Protocol | Total
Number analyzed (Participants) | 270 | 270 | 540
Number analyzed (ICUs) | 9 | 9 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: It doesn't the combined baseline and follow up equals the total of the participants to each arm
  years
    Baseline | 65.1 (15.5) | 63.4 (15.1) | 64.2 (15.3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: It doesn't the combined baseline and follow up equals the total of the participants to each arm
  Participants
    Baseline: Female | 113 | 100 | 213
    Baseline: Male | 157 | 170 | 327
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: ICUs]
  Canada | 4 | 5 | 9
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Prescribed Calories From Energy
Description: Total calories received from enteral nutrition/total prescription up to 12 evaluable ICU days
Time Frame: first 12 days
Population: This was a pre- post cluster RCT where the same 9 ICUs evaluated before and after randomization but the individuals at the ICUs are different. Some outcomes were analyzed at the ICU level while others were analyzed at the participant level. Ergo 522 is the total of 270 participants at baseline + 252 at follow up in the Pep up arm. Similarly in the standard feeding protocol 537= 270 at baseline + 267 at follow up
Measure: Mean (Standard Deviation); unit: percentage of prescription
Units Other Than Participants: ICUs
Arm/Group | PEP uP Protocol | Standard Feeding Protocol
Number analyzed (Participants) | 522 | 537
Number analyzed (ICUs) | 9 | 9
percentage of prescription
  Baseline time: number analyzed (Participants) | 270 | 270
  Baseline time | 32 (29.4) | 34.2 (30.9)
  Follow-up time: number analyzed (Participants) | 252 | 267
  Follow-up time | 43.6 (32.1) | 33.6 (29.5)

2. Secondary Outcome: Timeliness of Initiation of EN
Description: Time of the initiation of EN from ICU admit
Time Frame: 60 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Units Other Than Participants: ICUs
Arm/Group | PEP uP Protocol | Standard Feeding Protocol
Number analyzed (Participants) | 522 | 537
Number analyzed (ICUs) | 9 | 9
hours
  Baseline time: number analyzed (Participants) | 270 | 270
  Baseline time | 40.7 (30.6) | 33.6 (33.1)
  Follow-up time: number analyzed (Participants) | 252 | 267
  Follow-up time | 29.7 (31.4) | 35.2 (39.2)

3. Secondary Outcome: Percentage of Participants With Vomiting
Time Frame: 60 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PEP uP Protocol | Standard Feeding Protocol
Number analyzed (Participants) | 522 | 537
Participants
  Baseline time: number analyzed (Participants) | 270 | 270
  Baseline time | 12 | 20
  Follow-up time: number analyzed (Participants) | 252 | 267
  Follow-up time | 14 | 12

4. Secondary Outcome: Percentage of Participants With Pneumonia
Time Frame: 60 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | PEP uP Protocol | Standard Feeding Protocol
Number analyzed (Participants) | 522 | 537
Participants
  Baseline time: number analyzed (Participants) | 270 | 270
  Baseline time | 6 | 11
  Follow-up time: number analyzed (Participants) | 252 | 267
  Follow-up time | 7 | 16

5. Primary Outcome: Percentage of Prescribed Protein
Description: Total protein received from enteral nutrition/total prescription up to 12 evaluable ICU days
Time Frame: first 12 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of prescription
Units Other Than Participants: ICUs
Arm/Group | PEP uP Protocol | Standard Feeding Protocol
Number analyzed (Participants) | 522 | 537
Number analyzed (ICUs) | 9 | 9
percentage of prescription
  Baseline time: number analyzed (Participants) | 270 | 270
  Baseline time | 33.6 (31.1) | 34.2 (30.9)
  Follow-up time: number analyzed (Participants) | 252 | 267
  Follow-up time | 47.4 (34.7) | 33.6 (29.5)

ADVERSE EVENTS:
Time Frame: N/a not collected
Description: "0" Total Number of Participants at Risk (e.g.., serious and other [non-serious] adverse events were not collected or assessed as part of the study).
Arm/Group | PEP uP Protocol | Standard Feeding Protocol
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Sites struggled to embed the protocol in the initial admission order set and not able to achieve adequate dissemination of training materials. weekends or after hours, some patients admitted to the PEP uP sites did not actually receive the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No